CLINICAL TRIAL: NCT02694120
Title: Study on Complications, EfficAcy and Costs of Large Polypectomy
Acronym: SCALP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, MD, Valduce Hospital
Other Study IDs: 2016.2
Record Dates: First submitted 2016-01-29; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Polypectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

GROUPS / COHORTS (1):
- colonoscopy population

SUMMARY:
Colonoscopy has been shown to reduce the incidence and mortality of colorectal cancer, through the recognition and removal of pre-cancerous lesions, which in most cases evolve with a sequence that goes through formation of high-grade dysplasia (HGD).

The probability of HGD increases with the increase of the lesion of the polyp itself. Lesions> 2 cm are present in 1% of colonoscopy screening. The resection of these lesions presents a greater technical difficulty and consequently a decrease in the efficiency. The rate of incomplete resection reported in the literature reaches 10% while that of recurrence / residual adenoma 16.4 / 31.7%.

The aim of the study SCALP is to evaluate the incidence of complications, efficacy and cost of endoscopic resection of colic lesions> 2cm in a setting of clinical practice in an unselected population

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing large endoscopic polypectomy

Exclusion Criteria:

* pregnancy
* incapacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population undergoing large endoscopic polypectomy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
complications of large polypectomy | 15 days
  incidence of polypectomy-related adverse events

SECONDARY OUTCOMES:
costs of large polypectomy | 15 days
  assessment of the average cost per procedure, including devices and staff costs
efficacy of large polypectomy | 6 months
  assessment of residual adenoma at follow-up

REFERENCES:
- [Derived] Amato A, Radaelli F, Correale L, Di Giulio E, Buda A, Cennamo V, Fuccio L, Devani M, Tarantino O, Fiori G, De Nucci G, De Bellis M, Hassan C, Repici A; Bowell Group. Intra-procedural and delayed bleeding after resection of large colorectal lesions: The SCALP study. United European Gastroenterol J. 2019 Dec;7(10):1361-1372. doi: 10.1177/2050640619874176. Epub 2019 Sep 23. PMID 31839962